CLINICAL TRIAL: NCT07041528
Title: How Do Patients and Health Care Professionals Perceive De-implementation of Routine Follow-ups After Total Hip and Knee Arthroplasty? Protocol for a Nested Qualitative Study Within a Hybrid De-implementation Trial
Brief Title: Perceptions of De-implementing Routine Follow-ups After Hip and Knee Arthroplasty
Acronym: HAKA-QUALI
Status: Not yet recruiting | Type: Observational
Sponsor: Tergooi Medical Center (Other)
Collaborators: Reinier Haga Orthopedisch Centrum (Other); JointResearch (Other)
Responsible Party: Sponsor
Other Study IDs: N25.014; 10330042310003 (Other Grant/Funding Number: ZonMW)
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Hip Arthroplasty, Total; Knee Arthroplasty, Total
Keywords: Aftercare; Arthroplasty; Focus Groups; Hip; Interview [Publication Type]; Knee; Osteoarthritis; Patient Acceptance of Health Care; Qualitative Research
MeSH Terms: conditions — Osteoarthritis; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Routine Follow-up (RFU): Patients planned for total hip or knee surgery who will receive routinely scheduled follow-ups.
- Check-ups on-demand (COD): Patients planned for total hip or knee surgery who will receive check-ups on-demand.

SUMMARY:
After undergoing total hip or total knee arthroplasty, current guidelines recommend routine follow-up with an X-ray within 3 months and again at 1 year. Follow-up at 5 years (for hip arthroplasties) or every 5 years (for knee arthroplasties) is also considered worthwhile according to the guidelines. However, these follow-up appointments require considerable time from patients, caregivers, and healthcare professionals, and it is unclear whether they are truly beneficial. It is possible that a single follow-up within 3 months is sufficient. This could potentially prevent over 100,000 unnecessary hospital visits per year, resulting in significant cost savings. If patients or healthcare providers have concerns, they can always request an additional follow-up.

The HAKA trial consists of three different work packages (WPs).The quantitative work packages 1 (WP1) and 2 (WP2) will investigate the 1-year and 10-year follow-up. The qualitative third work package (WP3) will explore and compare the patients' and health care professionals' (HCPs) experiences with, and perceptions about, RFU and COD after total hip and knee arthroplasty. The aim of the overarching HAKA-trial is to safely reduce routine follow-up appointments after total hip or knee arthroplasty and to revise current clinical guidelines accordingly.

ELIGIBILITY:
Inclusion Criteria:

• A good command of the Dutch language

Exclusion Criteria:

* N/A

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients after total hip or knee arthroplasty who are enrolled in work package 1 or work package 2 of the main HAKA trial.
  * Health care professionals who have cared for at least 3 participants from the RFU or COD groups enrolled in work package 1 or work package 2 of the main HAKA trial.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
The participants' experiences with their follow-up regimen. | Experiences gained between the baseline clinical visit and a clinical visit one year later.
  The participants' experiences will be explored using a mix of semi-structured open-ended focus group questions.
The participants' satisfaction with their follow-up regimen. | Perceived satisfaction between the baseline clinical visit and a clinical visit one year later.
  The participants' satisfaction will be explored using a mix of semi-structured open-ended focus group questions.
The health care professionals' experiences with the different follow-up regimens. | Experiences gained between the baseline clinical visit and a clinical visit one year later.
  The health care professionals' experiences will be explored using a mix of semi-structured open-ended interview questions.
The health care professionals' satisfaction with the different follow-up regimens. | Perceived satisfaction between the baseline clinical visit and a clinical visit one year later.
  The health care professionals' satisfaction will be explored using a mix of semi-structured open-ended interview questions.
The participants' and health care professionals' acceptability of the two different follow-up regimens. | Acceptability of follow-up regimens from the baseline clinical visit to a clinical visit one year later.
  The participants' and health care professionals' acceptability of the two different follow-up regimens will be explored using a mix of semi-structured open-ended focus group questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Tergooi MC, Hilversum, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting data-including an overview of all themes, original Dutch quotes from focus groups and interviews, and their English translations-will be compiled in a table and made openly available via an online data repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning after publication with no end date.
Access Criteria: Anyone will be able to access the qualitative supportive data via an online data repository.

REFERENCES:
- [Background] Learmonth ID, Young C, Rorabeck C. The operation of the century: total hip replacement. Lancet. 2007 Oct 27;370(9597):1508-19. doi: 10.1016/S0140-6736(07)60457-7. PMID 17964352
- [Background] Price AJ, Alvand A, Troelsen A, Katz JN, Hooper G, Gray A, Carr A, Beard D. Knee replacement. Lancet. 2018 Nov 3;392(10158):1672-1682. doi: 10.1016/S0140-6736(18)32344-4. PMID 30496082
- [Background] Christensen M, Folkmar K. No clinical value of post-operative routine X-ray following uncomplicated cementless primary total hip arthroplasty. Dan Med J. 2013 Apr;60(4):A4613. PMID 23651720
- [Background] Hart AA, DeMik DE, Brown TS, Noiseux NO. Routine Radiographs After Total Joint Arthroplasty: Is There Clinical Value? J Arthroplasty. 2021 Jul;36(7):2431-2434. doi: 10.1016/j.arth.2021.02.050. Epub 2021 Feb 24. PMID 33714635
- [Background] Dargel J, Oppermann J, Bruggemann GP, Eysel P. Dislocation following total hip replacement. Dtsch Arztebl Int. 2014 Dec 22;111(51-52):884-90. doi: 10.3238/arztebl.2014.0884. PMID 25597367
- [Background] Blom AW, Beswick AD, Burston A, Carroll FE, Garfield K, Gooberman-Hill R, Harris S, Kunutsor SK, Lane A, Lenguerrand E, MacGowan A, Mallon C, Moore AJ, Noble S, Palmer CK, Rolfson O, Strange S, Whitehouse MR. Infection after total joint replacement of the hip and knee: research programme including the INFORM RCT [Internet]. Southampton (UK): National Institute for Health and Care Research; 2022 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK587029/ PMID 36469653
- [Background] Lindeque B, Hartman Z, Noshchenko A, Cruse M. Infection after primary total hip arthroplasty. Orthopedics. 2014 Apr;37(4):257-65. doi: 10.3928/01477447-20140401-08. PMID 24762833
- [Background] Schwartz AM, Farley KX, Guild GN, Bradbury TL Jr. Projections and Epidemiology of Revision Hip and Knee Arthroplasty in the United States to 2030. J Arthroplasty. 2020 Jun;35(6S):S79-S85. doi: 10.1016/j.arth.2020.02.030. Epub 2020 Feb 19. PMID 32151524
- [Background] Kunutsor SK, Barrett MC, Beswick AD, Judge A, Blom AW, Wylde V, Whitehouse MR. Risk factors for dislocation after primary total hip replacement: a systematic review and meta-analysis of 125 studies involving approximately five million hip replacements. Lancet Rheumatol. 2019 Oct;1(2):e111-e121. doi: 10.1016/S2665-9913(19)30045-1. Epub 2019 Sep 9. PMID 38229338
- [Background] Cassidy RS, O hEireamhoin S, Beverland DE. Guidelines for the follow-up of total hip arthroplasty: do they need to be revised? Bone Joint J. 2019 May;101-B(5):536-539. doi: 10.1302/0301-620X.101B5.BJJ-2018-0853.R2. PMID 31038998
- [Background] Lovelock TM, Broughton NS. Follow-up after arthroplasty of the hip and knee : are we over-servicing or under-caring? Bone Joint J. 2018 Jan;100-B(1):6-10. doi: 10.1302/0301-620X.100B1.BJJ-2017-0779.R1. PMID 29305444
- [Background] Smith LK, Dures E, Beswick AD. Systematic review of the clinical effectiveness for long-term follow-up of total hip arthroplasty. Orthop Res Rev. 2019 Jul 2;11:69-78. doi: 10.2147/ORR.S199183. eCollection 2019. PMID 31308766
- [Background] American Academy of Orthopaedic Surgeons. American Academy of Orthopaedic Surgeons Surgical Management of Osteoarthritis of the Knee Evidence-Based Clinical Practice Guideline. 2022
- [Background] Broughton N, Lovelock T, De Steiger R, Page R, Donnelly B, Solomon M, et al. Arthroplasty Society of Australia guidelines for long term follow-up of joint replacement patients. 2019
- [Background] Federatie Medisch Specialisten. Total hip prosthesis (THP). 2019
- [Background] ederatie Medisch Specialisten. Richtlijn Federatie Medisch Specialisten Totale Knieprothese (TKP). 2021
- [Background] Loppini M, Gambaro FM, Nelissen RGHH, Grappiolo G. Large variation in timing of follow-up visits after hip replacement: a review of the literature. EFORT Open Rev. 2022 Mar 17;7(3):200-205. doi: 10.1530/EOR-21-0016. PMID 35298395
- [Background] Kingsbury SR, Smith LK, Czoski Murray CJ, Pinedo-Villanueva R, Judge A, West R, Smith C, Wright JM, Arden NK, Thomas CM, Kolovos S, Shuweihdi F, Garriga C, Bitanihirwe BKY, Hill K, Matu J, Stone M, Conaghan PG. Safety of disinvestment in mid- to late-term follow-up post primary hip and knee replacement: the UK SAFE evidence synthesis and recommendations. Southampton (UK): National Institute for Health and Care Research; 2022 Jun. Available from http://www.ncbi.nlm.nih.gov/books/NBK581549/ PMID 35767667
- [Background] Matharu GS, Culliford DJ, Blom AW, Judge A. Projections for primary hip and knee replacement surgery up to the year 2060: an analysis based on data from The National Joint Registry for England, Wales, Northern Ireland and the Isle of Man. Ann R Coll Surg Engl. 2022 Jun;104(6):443-448. doi: 10.1308/rcsann.2021.0206. Epub 2021 Dec 23. PMID 34939832
- [Background] Inacio MCS, Paxton EW, Graves SE, Namba RS, Nemes S. Projected increase in total knee arthroplasty in the United States - an alternative projection model. Osteoarthritis Cartilage. 2017 Nov;25(11):1797-1803. doi: 10.1016/j.joca.2017.07.022. Epub 2017 Aug 8. PMID 28801208
- [Background] George J, Klika AK, Navale SM, Newman JM, Barsoum WK, Higuera CA. Obesity Epidemic: Is Its Impact on Total Joint Arthroplasty Underestimated? An Analysis of National Trends. Clin Orthop Relat Res. 2017 Jul;475(7):1798-1806. doi: 10.1007/s11999-016-5222-4. PMID 28054327
- [Background] Chen L, Zheng M, Chen Z, Peng Y, Jones C, Graves S, Chen P, Ruan R, Papadimitriou J, Carey-Smith R, Leys T, Mitchell C, Huang YG, Wood D, Bulsara M, Zheng MH. The burden of end-stage osteoarthritis in Australia: a population-based study on the incidence of total knee replacement attributable to overweight/obesity. Osteoarthritis Cartilage. 2022 Sep;30(9):1254-1262. doi: 10.1016/j.joca.2021.10.017. Epub 2021 Dec 7. PMID 34890810
- [Background] Smith LK. A survey of the current state of hip arthroplasty surveillance in the United Kingdom. Musculoskeletal Care. 2014 Dec;12(4):232-8. doi: 10.1002/msc.1077. Epub 2014 Jul 28. No abstract available. PMID 25065760
- [Background] Hacking C, Weinrauch P, Whitehouse SL, Crawford RW, Donnelly WJ. Is there a need for routine follow-up after primary total hip arthroplasty? ANZ J Surg. 2010 Oct;80(10):737-40. doi: 10.1111/j.1445-2197.2010.05346.x. PMID 21040336
- [Background] Kingsbury SR, Smith LKK, Pinedo-Villanueva R, Judge A, West R, Wright JM, Stone MH, Conaghan PG. Mid- to late-term follow-up of primary hip and knee arthroplasty: the UK SAFE evidence-based recommendations. Bone Jt Open. 2023 Feb 9;4(2):72-78. doi: 10.1302/2633-1462.42.BJO-2022-0149.R1. PMID 37051733
- [Background] National Joint Registry (NJR) Editorial Committee and contributors. 21st Annual Report, Hip Section. 2024.
- [Background] National Joint Registry (NJR) Editorial Committee and contributors. 21st Annual Report, Knee Section. 2024
- [Background] Pinedo-Villanueva R, Kolovos S, Burn E, Delmestri A, Smith LK, Judge A, Kingsbury SR, Stone MH, Conaghan PG. Association between outpatient follow-up and incidence of revision after knee and hip replacements: a population-based cohort study. BMC Musculoskelet Disord. 2023 Feb 8;24(1):106. doi: 10.1186/s12891-023-06190-7. PMID 36750857
- [Background] Schmitz PP, van Leent EAP, de Jong LD, van Susante JLC, Somford MP. The (un)necessity of regular postoperative follow-up of hemiarthroplasty for femoral neck fractures. Injury. 2021 Oct;52(10):2997-3001. doi: 10.1016/j.injury.2021.02.051. Epub 2021 Feb 26. PMID 33750587
- [Background] El Ashmawy AH, Dowson K, El-Bakoury A, Hosny HAH, Yarlagadda R, Keenan J. Effectiveness, Patient Satisfaction, and Cost Reduction of Virtual Joint Replacement Clinic Follow-Up of Hip and Knee Arthroplasty. J Arthroplasty. 2021 Mar;36(3):816-822.e1. doi: 10.1016/j.arth.2020.08.019. Epub 2020 Aug 15. PMID 32893060
- [Background] Richards JD, Stoddart M, Bolland B. Virtual Arthroplasty Follow-Up: Better for the Trust, Patients, and the Planet. Cureus. 2022 Nov 28;14(11):e31978. doi: 10.7759/cureus.31978. eCollection 2022 Nov. PMID 36589176
- [Background] Parkes RJ, Palmer J, Wingham J, Williams DH. Is virtual clinic follow-up of hip and knee joint replacement acceptable to patients and clinicians? A sequential mixed methods evaluation. BMJ Open Qual. 2019 Mar 1;8(1):e000502. doi: 10.1136/bmjoq-2018-000502. eCollection 2019. PMID 31259271
- [Background] Woolen SA, Kim CJ, Hernandez AM, Becker A, Martin AJ, Kuoy E, Pevec WC, Tutton S. Radiology Environmental Impact: What Is Known and How Can We Improve? Acad Radiol. 2023 Apr;30(4):625-630. doi: 10.1016/j.acra.2022.10.021. Epub 2022 Nov 16. PMID 36400705
- [Background] Zulman DM, Haverfield MC, Shaw JG, Brown-Johnson CG, Schwartz R, Tierney AA, Zionts DL, Safaeinili N, Fischer M, Thadaney Israni S, Asch SM, Verghese A. Practices to Foster Physician Presence and Connection With Patients in the Clinical Encounter. JAMA. 2020 Jan 7;323(1):70-81. doi: 10.1001/jama.2019.19003. PMID 31910284
- [Background] Healy P, McCrone L, Tully R, Flannery E, Flynn A, Cahir C, Arumugasamy M, Walsh T. Virtual outpatient clinic as an alternative to an actual clinic visit after surgical discharge: a randomised controlled trial. BMJ Qual Saf. 2019 Jan;28(1):24-31. doi: 10.1136/bmjqs-2018-008171. Epub 2018 Oct 5. PMID 30291181
- [Background] Abed H, Samson D, David M. Early Discharge and Patient-Initiated Follow-Up in Hand Surgery: A New Norm Following Simple Hand Surgery? Cureus. 2024 Jan 18;16(1):e52493. doi: 10.7759/cureus.52493. eCollection 2024 Jan. PMID 38371052
- [Background] Creswell J. Research Design: Qualitative, Quantitative and Mixed Methods Approaches. Third edition ed. Thousand Oaks, California: Sage Publications; 2022.
- [Background] Czoski Murray CJ, Kingsbury SR, Arden NK, Hewison J, Judge A, Matu J, O'Shea J, Pinedo-Villanueva R, Smith LK, Smith C, Thomas CM, West RM, Wright JM, Conaghan PG, Stone MH. Towards UK poSt Arthroplasty Follow-up rEcommendations (UK SAFE): protocol for an evaluation of the requirements for arthroplasty follow-up, and the production of consensus-based recommendations. BMJ Open. 2019 Jun 25;9(6):e031351. doi: 10.1136/bmjopen-2019-031351. PMID 31243039
- [Background] Yin R. Case Study Research and Applications. Design and Methods. 6th ed. Thousand Oaks, CA: SAGE Publications, Inc; 2018.
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Leask CF, Sandlund M, Skelton DA, Altenburg TM, Cardon G, Chinapaw MJM, De Bourdeaudhuij I, Verloigne M, Chastin SFM; GrandStand, Safe Step and Teenage Girls on the Move Research Groups. Framework, principles and recommendations for utilising participatory methodologies in the co-creation and evaluation of public health interventions. Res Involv Engagem. 2019 Jan 9;5:2. doi: 10.1186/s40900-018-0136-9. eCollection 2019. PMID 30652027
- [Background] Levitt HM, Motulsky SL, Wertz FJ, Morrow SL, Ponterotto JG. Recommendations for designing and reviewing qualitative research in psychology: Promoting methodological integrity. Qualitative Psychology. 2017;4(1):2-22. doi: 10.1037/qup0000082.
- [Background] Vasileiou K, Barnett J, Thorpe S, Young T. Characterising and justifying sample size sufficiency in interview-based studies: systematic analysis of qualitative health research over a 15-year period. BMC Med Res Methodol. 2018 Nov 21;18(1):148. doi: 10.1186/s12874-018-0594-7. PMID 30463515
- [Background] Waters S, Edmondston SJ, Yates PJ, Gucciardi DF. Identification of factors influencing patient satisfaction with orthopaedic outpatient clinic consultation: A qualitative study. Man Ther. 2016 Sep;25:48-55. doi: 10.1016/j.math.2016.05.334. Epub 2016 Jun 4. PMID 27422597
- [Background] Westbrook KW, Babakus E, Grant CC. Measuring patient-perceived hospital service quality: validity and managerial usefulness of HCAHPS scales. Health Mark Q. 2014;31(2):97-114. doi: 10.1080/07359683.2014.907114. PMID 24878401
- [Background] Wang Y, Liu C, Wang P. Patient satisfaction impact indicators from a psychosocial perspective. Front Public Health. 2023 Feb 22;11:1103819. doi: 10.3389/fpubh.2023.1103819. eCollection 2023. PMID 36908420
- [Background] Younis A, Elmubarak M, Elkhwad H, Baig MN, Saeed M, Omer A. Maximizing Satisfaction in Orthopedic Outpatient Clinics: Evidence From Ireland. Cureus. 2024 Jun 25;16(6):e63104. doi: 10.7759/cureus.63104. eCollection 2024 Jun. PMID 39055474
- [Background] Pollak KI, Alexander SC, Tulsky JA, Lyna P, Coffman CJ, Dolor RJ, Gulbrandsen P, Ostbye T. Physician empathy and listening: associations with patient satisfaction and autonomy. J Am Board Fam Med. 2011 Nov-Dec;24(6):665-72. doi: 10.3122/jabfm.2011.06.110025. PMID 22086809
- [Background] Dragovich A, Beltran T, Baylor GM, Swanson M, Plunkett A. Determinants of Patient Satisfaction in a Private Practice Pain Management Clinic. Pain Pract. 2017 Nov;17(8):1015-1022. doi: 10.1111/papr.12554. Epub 2017 Mar 3. PMID 28083999
- [Background] Chang CS, Chen SY, Lan YT. Service quality, trust, and patient satisfaction in interpersonal-based medical service encounters. BMC Health Serv Res. 2013 Jan 16;13:22. doi: 10.1186/1472-6963-13-22. PMID 23320786
- [Background] Kong MC, Camacho FT, Feldman SR, Anderson RT, Balkrishnan R. Correlates of patient satisfaction with physician visit: differences between elderly and non-elderly survey respondents. Health Qual Life Outcomes. 2007 Nov 24;5:62. doi: 10.1186/1477-7525-5-62. PMID 18036236
- [Background] Stephens AR, Rowberry TJ, Tyser AR, Kazmers NH. Evaluating opportunities for improved orthopedics outpatient satisfaction: an analysis of Press Ganey(R) Outpatient Medical Practice Survey responses. J Orthop Surg Res. 2020 Jan 28;15(1):28. doi: 10.1186/s13018-020-1567-1. PMID 31992339
- [Background] Sekhon M, Cartwright M, Francis JJ. Development of a theory-informed questionnaire to assess the acceptability of healthcare interventions. BMC Health Serv Res. 2022 Mar 1;22(1):279. doi: 10.1186/s12913-022-07577-3. PMID 35232455
- [Background] Hyman P. The Disappearance of the Primary Care Physical Examination-Losing Touch. JAMA Intern Med. 2020 Nov 1;180(11):1417-1418. doi: 10.1001/jamainternmed.2020.3546. No abstract available. PMID 32832987
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- See also: Published information about HAKA-trial work package 1 — https://www.zorgevaluatienederland.nl/evaluations/haka-1-year-fu
- See also: Published information about HAKA-trial work package 2 — https://www.zorgevaluatienederland.nl/evaluations/haka-10-year-fu